

## A Multi-Centre Prospective Randomised Control Trial to compare two articulating bearing surfaces, ceramic-on-metal and metalon-metal using 38 mm M2a acetabular cup, as used in cementless primary hip arthroplasty

**Protocol number: BMETEU.CR.EU11** 

NCT number: NCT00754520

COM vs. MOM



| Complete Protocol | A Multi-Centre Prospective Randomised Control Trial to compare two articulating bearing surfaces, ceramic-on-metal |
|---|---|
| Title | and metal-on-metal using 38 mm M2a acetabular cup, as used in cementless primary hip arthroplasty |
| Protocol Number | BMETEU.CR.EU11 |
| Short Protocol Title | COM vs MOM |
| Sponsor | Original: Biomet UK Ltd Administratively transferred: Biomet GSCC Administratively transferred: Zimmer GmbH, Zählerweg 4, 6300 Zug, Switzerland |
| Manufacturer | M2a-38 acetabular cup: Biomet Orthopaedics Inc, USA M2a-38 38 mm cobalt chromium molybdenum (CoCrMo) modular heads: Biomet Orthopaedics Inc, USA Biolox delta 38 mm ceramic femoral head: CeramTec AG now CeramTec GmbH, Germany |
| | Bi-Metric femoral stem: Biomet UK Limited, Bridgend, UK |
| Study Device(s) | COM articulation: M2a38 acetabular cup with ceramic head articulation Comparator: MOM articulation: M2a38 acetabular cup with metal head articualtion |
| Technical | |
| Documentation Reference Number | NA |
| | To evaluate the clinical outcome of the ceramic-on-metal (COM) articulation using M2a38 cup with metal-on-metal (MOM) articulation using the same cup. |
| | The metal ion release and additional cellular markers will be evaluated at predetermined postoperative intervals during the first 36 months. |
| Study | Primary objective |
| Objectives/Endpoints | The aim of the study is to demonstrate the non-inferiority of the ceramic-on-metal articulation using M2a-38 cup compared to the metal-on-metal articulation using the same cup in regards to the CCS rate at 2 year postoperative (delta = 10 % minimum clinically significant difference in rates). |
| | Each patient's CCS is defined as: |
| | Total Harris Hip Score ≥ 80 points, and |

COM vs. MOM



| | No acetabular or femoral revision or removal, and |
|---|---|
| | <ul> <li>No pending acetabular or femoral revision or removal as defined in radiographic evaluation by: <ul> <li>An acetabular radiographic assessment with all of the following: <ul> <li>Migration &lt; 4 mm, and</li> <li>Change in angle of inclination &lt; 4°, and</li> <li>Absence of osteolysis, and</li> <li>A femoral radiographic assessment with all of the following: <ul> <li>Subsidence &lt; 5 mm, and</li> <li>Absence of osteolysis.</li> <li>Absence of osteolysis.</li> </ul> </li> </ul> </li> </ul></li></ul> |
| | Secondary objective |
| | <ul> <li>Any reduction in metal ion release when using the ceramic-on-metal articulation compared to using metal-on-metal articulation.</li> <li>Harris Hip Score at each post-operative visit.</li> <li>Oxford Hip Score at each post-operative visit.</li> <li>Womac Score at each post-operative visit.</li> <li>Radiographic analysis at each post-operative visit.</li> <li>Complications (including revisions/removals).</li> <li>Long-term survivorship.</li> </ul> |
| Indications/Target Population | Patients suitable for primary Total Hip Replacement. |
| | Inclusion Criteria |
| | Patients suitable for primary Total Hip Replacement |
| | Patients with degenerative joint disease (inflammatory or non- |
| | inflammatory) or any of the composite diagnoses of: |
| | a. Osteoarthritis b. Avascular necrosis |
| | l b. Avascular necrosis |
| Inclusion/Exclusion | c. Legg Perthes |
| Inclusion/Exclusion<br>Criteria | c. Legg Perthes d. Rheumatoid Arthritis |
| • | c. Legg Perthes d. Rheumatoid Arthritis e. Diastrophic variant |
| • | c. Legg Perthes d. Rheumatoid Arthritis e. Diastrophic variant |
| • | c. Legg Perthes d. Rheumatoid Arthritis e. Diastrophic variant f. Fracture of the pelvis |
| | c. Legg Perthes d. Rheumatoid Arthritis e. Diastrophic variant f. Fracture of the pelvis g. Fused hip |

COM vs. MOM



| | Patients preoperative Harris Hip Score < 70 points |
|---|---|
| | Patients aged over 18 |
| | Patients with limited co-morbidity – ASA I – III |
| | Patients with normal urea and electrolyte levels and creatinine levels |
| | Patients must be able to understand instructions and be willing to return for follow-up |
| | Patients willing to provide blood and urine samples for metal ion analysis at follow-up |
| | Exclusion Criteria |
| | Patients preoperative Harris Hip Score > 70 points |
| | Pre-existing metal implants |
| | Patients with significant co-morbidity - ASA IV - V |
| | Dementia and inability to understand and follow instructions |
| | Neurological conditions affecting movement |
| | Pregnancy |
| | Presence of symptomatic arthritis in other lower limb joints |
| Study Design | Prospective Randomised Controlled Trial |
| | Group 1: Ø 38 mm metal femoral head articulating against Metal M2a-38 mm acetabular cup |
| | Group 2: |
| | Ø 38 mm ceramic femoral head articulating against Metal |
| | M2a-38 mm acetabular cup |
| Clinical Phase | Pre-market; COM articulation is not CE-marked |
| Sample Size | 300 planned, 150 per arm. |
| Janiple Size | 211 patients enrolled and included in study |
| Length of Study | 12 years (2 year enrollment, with a follow-up of 10 years) |
| Materials and<br>Methods | Case report forms will be completed either in-office or hospital at Pre-op, Surgery, Discharge, and the 6 week, 1-year, 2-year, and 5-year intervals. Case report forms will be completed at the 3-year, 7-year, and 10-year intervals either in-office, by phone or by mail. |
| Data Collection | Paper / electronic (Database: UK data in Access database; Finnish data in Joint Assist, study #339) |

COM vs. MOM



| Statistical Reporting | Data collected will be summarized and reported to each participating investigator. Statistical analysis will be conducted by Zimmer Biomet or its designee. Survivorship will be evaluated using Kaplan-Meier. |
|---|---|
| Scores/Performance Assessments | Harris Hip Score, Oxford Hip Score and WOMAC score |
| | The PMCF is compliant with the below: |
| Standards | <ul> <li>ISO 14155: 2020 - Clinical investigation of medical devices for human subjects - Good clinical practice.*</li> <li>The Declaration of Helsinki (DoH) - Ethical principles for medical research involving human subjects.</li> <li>(*) The study protocol was drafted according to another version of the ISO 14155. Adverse Event definitions and reporting are according to ISO 14155:2020.</li> </ul> |
| Study Funding | Funding for this clinical study is made available by Zimmer Biomet to support clinical data collection, IRB/EC review fees and other expenses associated with the conduct and execution of this study protocol as outlined in the fully executed Clinical Trial Agreement. |

## 1 STATISTICAL ANALYSIS PLAN

## 1.1 Sample Size

The sample size is determined by the primary end-point of composite clinical success (CCS) at two years post-operative. Since the aim is to demonstrate the non-inferiority of the COM compared to the MOM group in terms of CCS, the sample size calculation is based on the Blackwelder method<sup>[15]</sup>.

NULL hypothesis:  $p_2 - p_1 > \delta$ 

ALTERNATIVE hypothesis:  $p_2 - p_1 \le \delta$ 

 $\delta$  = 0.10 Difference in CCS rate between the MOM and COM groups that can

be considered clinically significant

Type I error ( $\alpha$ ): The error of rejecting Null hypothesis when it is actually true (false

positive)

COM vs. MOM



Type II error ( $\beta$ ): The error of failing to reject Null hypothesis when the alternative

hypothesis is true (false negative)

1.2

$$Z_{\alpha}$$
 = 1.645 When  $\alpha$  = 0.05

$$Z_{\beta}$$
 = 1.28 When  $\beta$  = 0.10, commonly used value in non-inferiority test

$$p_1 = 0.92$$
 Estimate CCS rate of COM group

$$p_2 = 0.92$$
 Estimate CCS rate of MOM group

Sample size required, N:

$$N = \frac{(Z_{\alpha} + Z_{\beta})^2 \big[ p_1 (1 - p_1) + p_2 (1 - p_2) \big]}{\delta^2}$$

$$N = \frac{(1.645 + 1.28)^2 [0.92(1 - 0.92) + 0.92(1 - 0.92)]}{0.10^2} = 126$$

Consider 7.5 % lost to follow-up per year, there will be 15 % cases lost to follow-up at 2 years post-operative.

$$\frac{126}{(1 - 0.15)} = 150$$
 Final sample size:

## 1.3 Statistical Analysis

Statistical Analysis of the results will be conducted using a suitable method by a qualified statistician.

COM vs. MOM